CLINICAL TRIAL: NCT02625909
Title: A Randomised Study of Interferon-free Treatment for Recently Acquired Hepatitis C in People Who Inject Drugs and People With HIV Coinfection.
Brief Title: Randomised Study of Interferon-free Treatment for Recently Acquired Hepatitis C in PWID and People With HIV Coinfection.
Acronym: REACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VHCRP1401
Record Dates: First submitted 2015-12-07; First posted 2015-12-09 (Estimated); Results first posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug: SOF/VEL for 6 weeks (Experimental): Open-label SOF/VEL 400mg/100mg co-formulated tablet once daily will be given to participants who are randomised into the short treatment duration arm (A) for 6 weeks.
  Interventions: Drug: SOF/VEL for 6 weeks
- Drug: SOF/VEL for 12 weeks (Experimental): Open-label SOF/VEL 400mg/100mg co-formulated tablet once daily will be given to participants who are randomised into the standard treatment duration arm (B) for 12 weeks.
  Interventions: Drug: SOF/VEL for 12 weeks

INTERVENTIONS:
Drug: SOF/VEL for 6 weeks — Open-label SOF/VEL 400mg/100mg once daily to be given to participants randomised to Arm A (6 weeks short treatment duration).
  Other Names: sofosbuvir (Sovaldi)/velpatasvir
  Arms: Drug: SOF/VEL for 6 weeks
Drug: SOF/VEL for 12 weeks — Open-label SOF/VEL 400mg/100mg once daily to be given to participants randomised to Arm B (12 weeks standard treatment duration).
  Other Names: sofosbuvir (Sovaldi)/velpatasvir
  Arms: Drug: SOF/VEL for 12 weeks

SUMMARY:
The aim of the study is to determine if treatment for recently acquired hepatitis C infection (with or without HIV coinfection) can be shortened when treating with the interferon-free therapy sofosbuvir/velpatasvir (SOF/VEL).

SOF/VEL is a new treatment for hepatitis C called direct acting antiviral which targets the hepatitis C virus replication cycle and has been shown in phase II studies in chronic HCV to be highly effective (SVR12 >95%) when given for 12 weeks.

Data has shown that treatment can be shortened when treating recently acquired HCV with interferon containing treatments. It is not known whether treatment with SOF/VEL can be shortened.

This study aims to find out if treatment for 6 weeks with open-label SOF/VEL is equivalent to treatment for 12 weeks with SOF/VEL in participants with recently acquired hepatitis C infection. The project is a randomised study where both participants and investigators would not find out the treatment duration of the participants until week 6 of treatment.

DETAILED DESCRIPTION:
Globally, 3-4 million new HCV infections are estimated to occur annually. People who inject drugs (PWID) represent one of the groups at highest risk of transmitting and acquiring infection with the majority of new (60%) and existing (80%) infections in developed countries occur in this population with HCV antibody prevalence estimated at 67% (60-80%). HIV-positive men-who-have-sex-with-men (MSM) are another high risk group for HCV acquisition.

Direct acting antivirals (DAA) has changed the treatment landscape for individuals with chronic HCV infection with interferon-free therapy offering high effectiveness and tolerability, even in "difficult-to-treat" populations.

Given the burden of HCV-related disease among PWID and HIV-positive MSM, strategies to enhance HCV assessment, treatment and prevention in these groups are urgently needed. Much of what is known about the timing of treatment initiation, regimen choice and duration of therapy in acute HCV infection comes from small observational studies and randomized controlled (randomly assigned into one or other of the different treatment groups)trials in selected populations with limited data on treatment in PWID and HIV co-infection. With recent rapid advances in HCV treatments, management strategies for acute HCV will evolve rapidly over the next few years.

The REACT study will compare the efficacy and safety of open-label SOF/VEL administered for 6 or 12 weeks in individuals with recent HCV infection. Participants will be randomised into receiving 6 weeks or 12 weeks treatment. Both investigators and participants will be blinded to the treatment duration until week 6 of treatment. The role and activity of DAA regimens in acute HCV infection requires evaluation, with the potential to be given as highly effective, short course interferon-sparing regimens, maximising acceptability to patients, encouraging uptake of treatment, limiting further transmission and preventing progression to chronic liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be eligible to participate in this study:

  1. Participants have voluntarily signed the informed consent form.
  2. 18 years of age or older.
  3. Detectable HCV RNA at screening (>10,000 IU/ml), and in the opinion of the investigator is unlikely to demonstrate spontaneous viral clearance
  4. HCV genotypes 1-6.
  5. HBsAg negative
  6. Compensated liver disease (Child-Pugh A)
  7. Negative pregnancy test at baseline (females of childbearing potential only).
  8. Medically stable on the basis of physical examination, medical history and vital signs
  9. Adequate English to provide reliable responses to the study questionnaires
  10. All fertile males and females must be using effective contraception during treatment and during the 30 days after treatment end.
  11. Recently acquired HCV infection (estimated duration of infection ≤12 months)*

Recently acquired HCV infection as defined by:

A) i) First anti-HCV Ab or HCV RNA positive within the previous 3 months and ii) Documented anti-HCV Ab negative within the 12 months prior to anti-HCV antibody positive result

OR

B) i) First anti-HCV Ab or HCV RNA positive within the previous 3 months and ii) Acute clinical hepatitis [jaundice or alanine aminotransferase (ALT)] > 10 X ULN) within the previous 6 months prior to first positive HCV antibody or HCV RNA, with no other cause of acute hepatitis identifiable

OR

C) For cases of recent HCV reinfection the following criteria are required:

Documented prior HCV antibody positive with HCV RNA negative on at least 2 occasions 6 months apart AND new HCV RNA positive within the previous 6 months

*Estimated duration of infection based on midpoint between last antibody negative or HCV RNA and first antibody positive or HCV RNA in the case of seroconversion and 6 weeks prior to date of maximum ALT in the case of acute hepatitis.

If co-infection with HIV is documented, the subject must meet the following criteria:

1. Antiretroviral (ARV) untreated for >8 weeks preceding screening visit with cluster of differentiation 4 (CD4) T cell count >500 cells/mm3 OR
2. On a stable ARV regimen for >8 weeks prior to screening visit, with CD4 T cell count >200 cells/mm3 and an undetectable plasma HIV RNA level.

   * Suitable ARV include:

     * Tenofovir (TDF) and tenofovir alafenamide (TAF)
     * Emtricitabine (FTC)
     * Rilpivirine
     * Dolutegravir
     * Elvitegravir/cobicistat
   * Contraindicated ARV include:

     * Efavirenz 50% reduction in velpatasvir (GS-5816) exposure
     * Didanosine
     * Zidovudine
     * Tipranavir Other ARV agents may be permissible at the time of study commencement pending further drug-drug interaction studies; please discuss with Study Principal Investigator.

Exclusion criteria:

Subjects who meet any of the exclusion criteria are not to be enrolled in this study.

1. History of any of the following:

   1. Clinically significant illness (other than HCV) or any other major medical disorder that may interfere with the participant treatment, assessment or compliance with the protocol; participants currently under evaluation for a potentially clinically significant illness (other than HCV) are also excluded.
   2. History of chronic pulmonary disease associated with functional limitation, severe cardiac disease, major organ transplantation or other evidence of severe illness, malignancy, or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
   3. Solid organ transplant
   4. Malignancy within 5 years prior to screening, with exception of specific cancers that may have been cured by surgical resection (basal cell skin cancer, etc.). Subjects under evaluation for possible malignancy are also excluded.
   5. Significant drug allergy (such as anaphylaxis or hepatotoxicity).
2. Subject shows evidence of significant liver disease in addition to hepatitis C, which may include but is not limited to drug- or alcohol-related cirrhosis, autoimmune hepatitis, hemochromatosis, Wilson's disease, non-alcoholic steatohepatitis (NASH), or primary biliary cirrhosis
3. Subject has known cirrhosis
4. Any of the following lab parameters at screening:

   1. Direct bilirubin > 1.5 x ULN
   2. Platelets < 50,000/μL
   3. Creatinine clearance (CLcr) < 60 mL/min
   4. Haemoglobin < 11 g/dL for females ; < 12 g/dL for males
   5. Albumin < 30g/L
5. Pregnant or nursing female.
6. Use of prohibited concomitant medications as described in section 5.2 in the protocol
7. Chronic use of systemically administered immunosuppressive agents (e.g. prednisone equivalent > 10 mg/day)
8. Known hypersensitivity to velpatasvir, sofosbuvir or formulation excipients.
9. Therapy with any anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) ≤6 months prior to the first dose of study drug.
10. Any investigational drug ≤6 weeks prior to the first dose of study drug.
11. Previous failure of therapy with sofosbuvir or an non-structural protein 5A (NS5A) inhibitor prior to the first dose of study drug.
12. Ongoing severe psychiatric disease as judged by the treating physician.
13. Frequent injecting drug use that is judged by the treating physician to compromise treatment safety.
14. Inability or unwillingness to provide informed consent or abide by the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail V Matthews, MbChB, PhD, Principal Investigator — The Kirby Institute, University of New South Wales Australia, Sydney, New South Wales, Australia, NSW 2052
Locations (25):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
- Australia (6):
  - Kirketon Road Centre, Sydney, New South Wales
  - St. Vincent's Hospital, Sydney, New South Wales
  - The Kirby Institute, University of New South Wales Australia, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
- Canada (4):
  - St Paul's Hospital, Vancouver, British Columbia
  - Cool Aid Community Health Centre, Victoria, British Columbia
  - Toronto General Hospital, Toronto, Ontario
  - Centre Hospitalier de l' Universite de Montreal, Montreal, Quebec
- Germany (4):
  - Praxis Dr Cordes, Berlin
  - Zentrum für Infektiologie Berlin-Prenzlauer Berg, Berlin
  - University Hospital of Bonn, Bonn
  - Infektio-Research GmbH, Frankfurt
- Academic Medical Centre, University of Amsterdam, Amsterdam, Netherlands
- Auckland City Hospital, Auckland, New Zealand
- Switzerland (3):
  - University Hospital Zurich, Zurich, Canton of Zurich
  - Bern University Hospital, Bern
  - Fondazione Epatocentro Ticino, Lugano
- United Kingdom (4):
  - Brighton & Sussex University Hospitals NHS Trust, Brighton, Brigton and Hove
  - Pennine Acute Hospitals NHS Trust, Manchester, Lancashire
  - Royal Free Hospital, London
  - Chelsea & Westminster Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
No individual participant data will be shared. The results of the project will be presented at scientific meetings, and published in peer reviewed scientific literature. Sharing of data generated by this project is an essential part of our proposed activities and will be carried out in several different ways. We plan to make our results available to the community of scientists interested in recently acquired hepatitis C, community organisations representing the affected communities and participants. We also welcome collaboration with others who could make use of data and samples.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Available following publication of the primary manuscript, indefinitely
Access Criteria: Submission of a research concept sheet proposal to the study Principal Investigator for review and approval by the protocol steering committee,

REFERENCES:
- [Derived] Carson JM, Barbieri S, Cunningham E, Mao E, van der Valk M, Rockstroh JK, Hellard M, Kim A, Bhagani S, Feld JJ, Gane E, Thurnheer MC, Bruneau J, Tu E, Dore GJ, Matthews GV, Martinello M; REACT study group. Sexual and drug use risk behaviour trajectories among people treated for recent HCV infection: the REACT study. J Int AIDS Soc. 2023 Sep;26(9):e26168. doi: 10.1002/jia2.26168. PMID 37675828
- [Derived] Matthews GV, Bhagani S, Van der Valk M, Rockstroh J, Feld JJ, Rauch A, Thurnheer C, Bruneau J, Kim A, Hellard M, Shaw D, Gane E, Nelson M, Ingiliz P, Applegate TL, Grebely J, Marks P, Martinello M, Petoumenos K, Dore GJ; REACT study group; Protocol Steering Committee; Coordinating Centre; Site Principal Investigators. Sofosbuvir/velpatasvir for 12 vs. 6 weeks for the treatment of recently acquired hepatitis C infection. J Hepatol. 2021 Oct;75(4):829-839. doi: 10.1016/j.jhep.2021.04.056. Epub 2021 May 21. PMID 34023350

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total 277 participants screened for protocol eligibility. Of 277 participants, 55 participants did not meet the protocol eligibility and excluded. Hence, a total 222 participants were enrolled into the study.
Pre-assignment Details: Of 277 participants screened for eligibility,55 were excluded [not meeting inclusion criteria (n=38),consent withdrawn/refusal (n=7),lost to follow-up (n=4), other (n=6)] and 26 commenced treatment but not randomized were excluded [between baseline (BSL) and wk 6 at Data Safety & Monitoring Board (DSMB) advice (n=9),in screening at DSMB advice (n=12),lost to follow-up before wk 6 (n=5)]. 196 were randomized with 8 (4 in each arm) excluded following DSMB advice,hence a final population of 188.
Groups:
- Drug: Sofosbuvir/Velpatasvir (SOF/VEL) for 6 Weeks: Open-label sofosbuvir/velpatasvir (SOF/VEL) 400mg/100mg co-formulated tablet once daily will be given to participants who are randomised into the short treatment duration arm (A) for 6 weeks.
  SOF/VEL for 6 weeks: Open-label SOF/VEL 400mg/100mg once daily to be given to participants randomised to Arm A (6 weeks short treatment duration).
- Drug: Sofosbuvir/Velpatasvir (SOF/VEL) for 12 Weeks: Open-label sofosbuvir/velpatasvir (SOF/VEL) 400mg/100mg co-formulated tablet once daily will be given to participants who are randomised into the standard treatment duration arm (B) for 12 weeks.
  SOF/VEL for 12 weeks: Open-label SOF/VEL 400mg/100mg once daily to be given to participants randomised to Arm B (12 weeks standard treatment duration).
Period: Overall Study
Arm/Group | Drug: Sofosbuvir/Velpatasvir (SOF/VEL) for 6 Weeks | Drug: Sofosbuvir/Velpatasvir (SOF/VEL) for 12 Weeks
Started | 93 | 95
Completed | 76 | 86
Not Completed | 17 | 9
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 3 | 5
Not completed — Lack of Efficacy | 9 | 2
Not completed — Reinfection | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug: Sofosbuvir/Velpatasvir (SOF/VEL) for 6 Weeks | Drug: Sofosbuvir/Velpatasvir (SOF/VEL) for 12 Weeks | Total
Number analyzed (Participants) | 93 | 95 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (10.3) | 43.4 (10.2) | 43.8 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 91 | 91 | 182
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/White | 79 | 78 | 157
  Asian | 4 | 4 | 8
  Black or African American | 0 | 2 | 2
  Other | 9 | 8 | 17
  Unknown or not reported | 1 | 3 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 8 | 11
  Not Hispanic or Latino | 89 | 87 | 176
  Unknown or not reported | 1 | 0 | 1
Type of hepatitis C virus (HCV) infection [Count of Participants; unit: Participants]
  Primary infection | 59 | 60 | 119
  Reinfection | 34 | 35 | 69
Human Immunodeficiency Virus (HIV) positive [Count of Participants; unit: Participants] | 65 | 65 | 130
Baseline HCV ribonucleic acid (RNA) [Median (Inter-Quartile Range); unit: log10 IU/ml] | 5.6 [4.8 to 6.5] | 5.4 [4.3 to 6.3] | 5.6 [4.6 to 6.5]
HCV genotype [Count of Participants; unit: Participants]
  1a | 58 | 57 | 115
  1b | 4 | 2 | 6
  1 unknown subtype | 1 | 0 | 1
  2 | 0 | 4 | 4
  3 | 15 | 17 | 32
  4 | 15 | 15 | 30
Mode of HCV exposure [Count of Participants; unit: Participants]
  Injecting drug use | 18 | 22 | 40
  Sexual exposure with person(s) of opposite sex | 3 | 4 | 7
  Sexual exposure with person(s) of same sex | 69 | 66 | 135
  Occupational (needle stick or other exposure) | 0 | 1 | 1
  Use of non-injectable recreational drugs | 1 | 0 | 1
  Other | 2 | 2 | 4
Max alanine aminotransferase (ALT) [Median (Inter-Quartile Range); unit: International units per liter (IU/L)] | 364 [152 to 799] | 360 [155 to 871] | 362 [154 to 847]
Baseline ALT [Median (Inter-Quartile Range); unit: International units per liter (IU/L)] | 114 [56 to 257] | 128 [69 to 222] | 126 [62 to 250]
Symptomatic presentation [Count of Participants; unit: Participants] | 16 | 14 | 30
Estimated duration of infection to baseline [Median (Inter-Quartile Range); unit: weeks] | 26.1 [17 to 33.8] | 25.0 [17 to 35.4] | 25.8 [17 to 35.2]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Undetectable HCV RNA at 12 Weeks Post End of Treatment (SVR12) Following SOF/VEL for 6 Weeks as Compared With 12 Weeks in People With Recent HCV Infection- Among Intention-to-treat (ITT) Population
Description: To evaluate the proportion of participants with HCV RNA below the level of quantification at 12 weeks post treatment following SOF/VEL for 6 weeks as compared with 12 weeks in people with recent HCV infection- among intention-to-treat (ITT) population The ITT population included all randomized participants, with loss to follow-up deemed treatment failure.
Time Frame: 12 weeks post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Drug: SOF/VEL for 6 Weeks | Drug: SOF/VEL for 12 Weeks
Number analyzed (Participants) | 93 | 95
Participants | 76 | 86

2. Secondary Outcome: Number of Participants With Undetectable HCV RNA at 12 Weeks Post End of Treatment (SVR12) Following SOF/VEL for 6 Weeks as Compared With 12 Weeks in People With Recent HCV Infection- Among Modified Intention-to-treat (ITT) Population
Description: To evaluate the proportion of participants with HCV RNA below the level of quantification at 12 weeks post treatment following SOF/VEL for 6 weeks as compared with 12 weeks in people with recent HCV infection- among modified intention-to-treat (ITT) population The modified ITT population included participants in the ITT population, but excluded those with non-virological reasons for treatment failure (including death and loss to follow-up) and reinfection.
Time Frame: 12 Weeks Post End of Treatment
Population: The modified ITT population included participants in the ITT population, but excluded those with non-virological reasons for treatment failure (including death and loss to follow-up) and reinfection. 8 out of 93 individuals in short arm (3 reinfections, 2 deaths and 3 lost to follow ups) and 7 out of 95 individuals in standard arm (2 reinfections and 5 lost to follow ups) were excluded. Therefore the final number for analysis population were 85 and 88 in short and standard arm, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug: SOF/VEL for 6 Weeks | Drug: SOF/VEL for 12 Weeks
Number analyzed (Participants) | 85 | 88
Participants | 76 | 86

3. Secondary Outcome: Number of Participants With Undetectable HCV RNA at End of Treatment (ETR) of SOF/VEL for 6 Weeks as Compared With 12 Weeks in People With Recent HCV Infection- Among Intention-to-treat (ITT) Population
Description: To evaluate the proportion of participants with HCV RNA below the level of quantification at end of treatment of SOF/VEL for 6 Weeks as compared With 12 Weeks in People With Recent HCV Infection The ITT population included all randomized participants, with loss to follow-up deemed treatment failure.
Time Frame: End of treatment - week 6 of the shortened treatment duration arm, and week 12 of the standard treatment duration arm
Measure: Count of Participants; unit: Participants
Arm/Group | Drug: SOF/VEL for 6 Weeks | Drug: SOF/VEL for 12 Weeks
Number analyzed (Participants) | 93 | 95
Participants | 85 | 87

4. Secondary Outcome: Number of Participants With Undetectable HCV RNA at 12 Weeks Post End of Treatment (SVR12) Following SOF/VEL for 6 Weeks as Compared With 12 Weeks in People With Recent HCV Infection- Among Per Protocol (PP) Population
Description: To evaluate the proportion of participants with HCV RNA below the level of quantification at 12 weeks post treatment following SOF/VEL for 6 weeks as compared with 12 weeks in people with recent HCV infection- among Per Protocol (PP) population The per protocol population included participants who received >90% of scheduled treatment for >90% of the scheduled treatment period with follow-up virologic data at SVR12 (excluding reinfection and retreatments)
Time Frame: 12 weeks post treatment
Population: The per protocol population included participants who received >90% of scheduled treatment for >90% of the scheduled treatment period with follow-up virologic data at SVR12 (excluding reinfection and retreatments) which was 74 and 77 for short and standard arm, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug: SOF/VEL for 6 Weeks | Drug: SOF/VEL for 12 Weeks
Number analyzed (Participants) | 74 | 77
Participants | 69 | 77

ADVERSE EVENTS:
Time Frame: All adverse events up to 4 weeks after the last dose of study drug administration, an average of 10 weeks (arm A) and 16 weeks (arm B).
Arm/Group | Drug: SOF/VEL for 6 Weeks | Drug: SOF/VEL for 12 Weeks
All-Cause Mortality (participants affected / at risk) | 2/93 | 0/95
Serious Adverse Events (participants affected / at risk) | 1/93 | 5/95
Other Adverse Events (participants affected / at risk) | 34/93 | 48/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Drug: SOF/VEL for 6 Weeks (N=93) | Drug: SOF/VEL for 12 Weeks (N=95)
Drug withdrawal syndrome (General disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Opium addiction (Psychiatric disorders) | 0 | 1 — Drug dependence
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Cellulitis of leg (Infections and infestations) | 0 | 1 — Cellulitis
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Drug: SOF/VEL for 6 Weeks (N=93) | Drug: SOF/VEL for 12 Weeks (N=95)
Fatigue (General disorders) | 9 | 12
Headache (Nervous system disorders) | 6 | 11
Nasopharyngitis (Infections and infestations) | 8 | 9
Nausea (Gastrointestinal disorders) | 5 | 9
Diarrhoea (Gastrointestinal disorders) | 6 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-06-04): https://cdn.clinicaltrials.gov/large-docs/09/NCT02625909/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT02625909/SAP_001.pdf